CLINICAL TRIAL: NCT07278323
Title: Hormone Replacement Therapy as an Adjunct Treatment for Adhesive Capsulitis of the Shoulder (Frozen Shoulder) in Peri- and Postmenopausal Women
Brief Title: Frozen Shoulder and Hormone Replacement Therapy
Acronym: FSHRT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-44965
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis of the Shoulder; Frozen Shoulder
Keywords: Frozen Shoulder; Hormone Replacement Therapy; Perimenopause
MeSH Terms: conditions — Bursitis | interventions — Hormone Replacement Therapy; Adrenal Cortex Hormones; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hormone Replacement Therapy plus standard care (Experimental): Participants will be prescribed HRT for 6 months (estrogen patch and oral progestin) in addition to receiving a steroid injection at the shoulder and referral to physical therapy.
  Interventions: Drug: Hormone Replacement Therapy (HRT); Drug: Corticosteroid and 1%lidocain; Behavioral: physical therapy
- Standard Care (Active Comparator): Participants will receive standard care for frozen shoulder including a steroid injection at the shoulder and referral to physical therapy
  Interventions: Drug: Corticosteroid and 1%lidocain; Behavioral: physical therapy

INTERVENTIONS:
Drug: Hormone Replacement Therapy (HRT) — Participants will receive HRT for 6 months consisting of 0.5mg estradiol skin patch and 100mg of oral daily progestin
  Arms: Hormone Replacement Therapy plus standard care
Drug: Corticosteroid and 1%lidocain — Ultrasound-guided glenohumeral joint injections will be performed in clinic by a board-certified fellowship-trained primary care sports medicine physician with expertise performing ultrasound-guided joint injections. Injections will be performed using standard aseptic technique after obtaining informed consent. For local anesthesia, 1 mL of 1% lidocaine will be injected with a 25 gauge 2-inch needle into the skin and subcutaneous tissues. Following this, a 22 gauge 2.5-inch needle will be used to inject a 5 mL combination of 1 mL of 40 mg/mL triamcinolone, 2 mL of 0.2% ropivacaine, and 2 mL of normal saline into the glenohumeral joint.
Behavioral: physical therapy — Patients will be referred to physical therapy to complete on their own and will be given an at home program to follow while they wait to see therapists.

SUMMARY:
The purpose of this study is to determine the effects of hormone replacement therapy (HRT) in addition to standard treatment on frozen shoulder symptoms in women with age-related changes to their menstrual cycle. Frozen shoulder refers to the condition a doctor diagnosed the participant with regarding shoulder pain, stiffness, and progressive loss of range of motion. Age-related menstrual cycle changes, known as perimenopause and/or menopause, refers to a change or stoppage of monthly menstrual cycles. Other symptoms participants may be experiencing include vaginal dryness, hot flashes, or night sweats. Hormone replacement therapy (HRT) refers to medicine with female hormones in it. For this study, HRT will be in the form of a patch that goes on the skin and a daily oral pill. Participants will be randomly assigned to receive either HRT plus standard care, or only standard care. Follow-up tests will be completed at 6 months of treatment to assess participant progress.

DETAILED DESCRIPTION:
Adhesive capsulitis of the shoulder (ACS), also known as frozen shoulder, affects up to 5% of the population with most cases occurring in peri- and postmenopausal women. This condition is debilitating, negatively impacting quality of life, yet current treatments are insufficient. There are mechanistic studies and biological plausibility to suggest the onset of this condition is associated with hormonal involvement, specifically estrogen. Given hormone replacement therapy (HRT) is widely prescribed to women experiencing menopause-related symptoms, investigators propose using HRT as an adjunct treatment for ACS. The primary objective of this study is to evaluate patient-reported outcomes using the American Shoulder and Elbow Surgeons (ASES) score following treatment with HRT + standard care versus standard care alone. The secondary objective is to determine changes in range of motion (ROM) and functional workspace using both routine clinical metrics and a novel clinical marker-less movement analysis system. Investigators hypothesize that HRT can improve pain scores and ROM limitations in peri- and postmenopausal women who present with ACS. Investigators will recruit 60 women who are peri- or postmenopausal and employ a longitudinal randomized controlled trial to determine the effects of HRT + standard treatment on ACS symptom severity. All participants will receive standard care of physical therapy and a glenohumeral joint steroid injection; the experimental group will also receive HRT. Measures will be repeated after six months of treatments. Within- and between-group changes in pain scores, ROM, and functional workspace will be evaluated using repeated measures ANOVAs with Tukey's multiple comparisons test as indicated by treatment groups. An alpha level of 0.05 will be used to determine statistical significance for all measures. This pilot project will provide critical preliminary data to support future extramural funding applications to government agencies, foundations, and industry partners.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adhesive capsulitis of the shoulder

Exclusion Criteria:

* History of hormone sensitive cancer
* Bilateral adhesive capsulitis of the shoulder
* Currently using hormonal treatments including contraceptives

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients are eligible
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Function Scores | 6 months
  Pain in affected shoulder measured on the American Shoulder and Elbow Surgeons (ASES) shoulder function scale. Scores range from 0 to 100 with 0 indicating the lowest level of shoulder function and 100 indicating the highest level of shoulder function.
Shoulder range of motion via goniometry measures. | 6 months
  Investigators will assess the degree of flexion, extension, adduction, and abduction in the shoulder to determine range of motion.

OTHER OUTCOMES:
Shoulder Functional Workspace | 6 months
  Kinectigram by Bioniks will be used to evaluate the functional workspace of the shoulder. This motion capture system assesses the ability of participants to reach with their hands to determine the total area the hand can reach relative to the shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Wong, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopaedic Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klair JS, Yang JD, Abdelmalek MF, Guy CD, Gill RM, Yates K, Unalp-Arida A, Lavine JE, Clark JM, Diehl AM, Suzuki A; Nonalcoholic Steatohepatitis Clinical Research Network. A longer duration of estrogen deficiency increases fibrosis risk among postmenopausal women with nonalcoholic fatty liver disease. Hepatology. 2016 Jul;64(1):85-91. doi: 10.1002/hep.28514. Epub 2016 Apr 5. PMID 26919573
- [Background] Hamed-Hamed D, Rodriguez-Perez C, Pruimboom L, Navarro-Ledesma S. Influence of the metabolic and inflammatory profile in patients with frozen shoulder - systematic review and meta-analysis. BMC Musculoskelet Disord. 2025 May 15;26(1):475. doi: 10.1186/s12891-025-08706-9. PMID 40375116
- [Background] Kraal T, Lubbers J, van den Bekerom MPJ, Alessie J, van Kooyk Y, Eygendaal D, Koorevaar RCT. The puzzling pathophysiology of frozen shoulders - a scoping review. J Exp Orthop. 2020 Nov 18;7(1):91. doi: 10.1186/s40634-020-00307-w. PMID 33205235
- [Background] Cogan CJ, Cevallos N, Freshman RD, Lansdown D, Feeley BT, Zhang AL. Evaluating Utilization Trends in Adhesive Capsulitis of the Shoulder: A Retrospective Cohort Analysis of a Large Database. Orthop J Sports Med. 2022 Jan 25;10(1):23259671211069577. doi: 10.1177/23259671211069577. eCollection 2022 Jan. PMID 35097146